CLINICAL TRIAL: NCT00029159
Title: The Effects of Androgen, Estrogen, and the Combination of Androgen and Estrogen on Growth Rate and Cognitive Function of Growth Hormone-treated Girls With Turner Syndrome
Brief Title: The Effect of Androgen and Growth Hormone on Height and Learning in Girls With Turner Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NS032531 (NIH)
Record Dates: First submitted 2002-01-08; First posted 2002-01-09 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Turner Syndrome
Keywords: Turner syndrome; estrogen; androgen; growth hormone
MeSH Terms: conditions — Turner Syndrome | interventions — Estrogens; Androgens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: estrogen; Drug: androgen
- 2 (Placebo Comparator)
  Interventions: Drug: estrogen; Other: placebo

INTERVENTIONS:
Drug: estrogen — Participants were started on ethinyl estradiol at a daily dose of 50ng/kg at the beginning of the 3rd year of the study. The estrogen was continued until study end.
Drug: androgen — Oxandrolone or placebo capsule, .06mg/kg/day, orally, for 2 years
  Arms: 1
Other: placebo — an inactive substance
  Arms: 2

SUMMARY:
The purposes of this study are to learn whether treatment with an androgen type hormone will improve the visual-spatial problems associated with Turner syndrome, and to evaluate the effect growth hormone, with and without androgen, has on growth.

DETAILED DESCRIPTION:
Turner syndrome is associated with short stature, multiple physical stigmata, absent pubertal development, and increased learning problems. This study is designed to (1) examine the effects of sex steroids (androgen and estrogen) on multiple variables including growth rate, GH binding protein, IGF-I, IGFBP3, and cognitive function in the setting of supplemental growth hormone administration and (2) to investigate any synergistic or additive effects of the androgen and estrogen combination versus each alone, on the above variables.

ELIGIBILITY:
* Karyotype diagnosis compatible with Turner syndrome, but no presence of any Y material in the peripheral karyotype unless a gonadectomy has been performed;
* Chronological age between 10.0 and 14.9 years;
* Bone age less than or equal to 12 years; and
* No treatment with estrogen, androgen, growth hormone, or any other growth-promoting agents exceeding 12 months, and no treatment with any of these agents in the previous 3 months.

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 1992-11; Primary Completion 2007-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cognitive function in girls with Turner Syndrome | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Judith L. Ross, M.D., Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - National Institutes of Health, Bethesda, Maryland
  - Thomas Jefferson University Hospital, 1025 Walnut Street, Suite 726, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Zeger MP, Shah K, Kowal K, Cutler GB Jr, Kushner H, Ross JL. Prospective study confirms oxandrolone-associated improvement in height in growth hormone-treated adolescent girls with Turner syndrome. Horm Res Paediatr. 2011;75(1):38-46. doi: 10.1159/000317529. Epub 2010 Aug 20. PMID 20733274